CLINICAL TRIAL: NCT02260713
Title: Autologous Bone Marrow Cell Transplantation in Persons With Acute Spinal Cord Injury- An Indian Pilot Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indian Spinal Injuries Centre (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISIC-BMC
Record Dates: First submitted 2014-09-16; First posted 2014-10-09 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2016-02

CONDITIONS: Acute Spinal Cord Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): control subjects with acute complete spinal cord injury who would not receive any bone marrow transplantation.
- Transplantation via intrathecal route (Experimental): Subjects with acute complete spinal cord injury who receive autologous bone marrow cell transplantation via lumber puncture
  Interventions: Biological: autologous bone marrow cell
- Transplantation via intralesional route (Experimental): Subjects with acute complete spinal cord injury who receive autologous bone marrow cell transplantation via durotomy and injection at the lesional site .
  Interventions: Biological: autologous bone marrow cell

INTERVENTIONS:
Biological: autologous bone marrow cell — Transplantation of 200 million cells in 1.8 ml of autologous plasma in a single sitting. In case of intralesional route, the cells were delivered in one sitting at six sites ( 2 above the lesion, 2 at the lesion and 2 below the lesion) as 0.3 ml aliquots each. In case of Intrathecal route, the cells were delivered as a single injection of 1.8ml via lumbar puncture.
  Arms: Transplantation via intralesional route; Transplantation via intrathecal route

SUMMARY:
Pilot study on 7 subjects in each group (total 21 subjects) to establish the safety and feasibility of autologous bone marrow cell transplantation in case of acute complete spinal cord injury by each of the following techniques and a corresponding number of controlled subjects:

* Directly into the injured site with a syringe after exposing the spinal cord.
* By Intrathecal injection.

DETAILED DESCRIPTION:
Intervention : Autologous bone marrow cell: Transplantation of the autologous bone marrow cell transplantation through one of the below mentioned techniques: 1. Directly into the injured spinal cord site with a syringe after exposing the spinal cord. 2. By Intrathecal injection. Number of cells Injected: 200 million cells in 1.8 ml of autologous plasma. In case of Direct delivery, the cells were delivered in one sitting at six sites ( 2 above the lesion, 2 at the lesion and 2 below the lesion) as 0.3 ml aliquots each. In case of Intrathecal injection, the cells were delivered as a single injection of 1.8ml via lumbar puncture. Frequency of Injection: Single Total duration of Therapy: The procedure of Bone marrow harvesting, enrichment and transplantation was completed in a single setting of approximately 2-3 hours. The transplantation procedure in case of Direct delivery took 2 mins per injection site that is approximately 12 mins and in case of lumbar puncture the transplantation procedure took approximately 2 mins.

Comparator Agent:Control: control subjects with acute complete spinal cord injury who would not receive any bone marrow transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Acute spinal cord injury between 10 days and 14 days post injury.
2. The subject must have a traumatic spinal cord injury between the spinal segmental levels T1 and T12 (Neurological Level).
3. Must have a complete injury (ASIA-A).

Exclusion Criteria:

1. Subject whose medical condition requires mechanical ventilation.
2. Subjects with neurological level of injury above T1 and below T12.
3. Subjects more than 14 days and less than 10 days post-injury.
4. Lower motor neuron injury.
5. Subjects with pathological fracture.
6. Spinal Injuries in subjects with Ankylosing Spondylitis.
7. Subjects with extremes of age: less than 18 years or more than 50 years.
8. Subjects with pre-existing severe medical disease which would affect the outcome like severe diabetes, rheumatoid arthritis.
9. Subjects with Psychological disorders.
10. Female subjects with pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Examine for improvement in the ASIA classification. | up to 5 years
  Blinded assessors will examine for improvement in the ASIA classification of at least one grade by 12 months or change from baseline of 10 points or more in total motor score, with consideration of their distribution along the neuraxis, from the ASIA Impairment Scale (AIS) manual motor test by 12 months.

SECONDARY OUTCOMES:
Any voluntary movement by additional muscle groups not included in International Standards for Neurological Classification of Spinal Cord Injury | up to 5 years
Improvement by at least 1 point on the WISCI scale | up to 5 years
Decrease in spasticity by one grade or more as assessed by Modified Ashworth Spasticity Scale | up to 5 years
Improvement in ASIA sensory examination | up to 5 years
Improvements in SCIM score | up to 5 years
Psychological evaluation | up to 5 years
Improvements in EMG | up to 5 years
Improvements in SSEP | up to 5 years
Improvements in MEP | up to 5 years
Significant change in any of the variables included in urodynamic assessment | up to 5 years
Improvements in any of the variables included in ISCIS | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr Harvinder S Chhabra, MS, Principal Investigator — Indian Spinal Injuries Centre
Locations (1):
- Indian Spinal Injury Center, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chhabra HS, Sarda K, Arora M, Sharawat R, Singh V, Nanda A, Sangodimath GM, Tandon V. Autologous bone marrow cell transplantation in acute spinal cord injury--an Indian pilot study. Spinal Cord. 2016 Jan;54(1):57-64. doi: 10.1038/sc.2015.134. Epub 2015 Aug 18. PMID 26282492